CLINICAL TRIAL: NCT01515332
Title: Energy Expenditure Methodology
Status: Completed | Type: Observational
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 131306
Record Dates: First submitted 2011-11-23; First posted 2012-01-24 (Estimated); Last update posted 2015-09-10 (Estimated); Status verified 2015-09

CONDITIONS: Healthy Adults

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is simply to test the repeatability of the indirect calorimetry instrument the investigators use for our clinical studies.

DETAILED DESCRIPTION:
Participants will be required to attend two study visits at the Arkansas Children's Nutrition Center. During the first visit, informed consent will be obtained, participant will be measured and an indirect calorimetry assessment to measure resting energy expenditure will be performed. During the second visit, we will repeat the indirect calorimetry assessment to measure resting energy expenditure.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older

Exclusion Criteria:

* pulmonary or respiratory disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy adults from the surrounding community
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2011-03; Primary Completion 2011-03 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
repeatability of test results | 2-3 hours up to 2-3 days
  test the repeatability of the indirect calorimetry instrument used in other clinical studies at our center

CONTACTS AND LOCATIONS:
Locations (1):
- Arkansas Children's Nutrition Center, Little Rock, Arkansas, United States